CLINICAL TRIAL: NCT00200538
Title: Double-blind, Parallel Group, Placebo-controlled Trial of the Efficacy and Tolerability of Memantine (20 mg) in Frontotemporal Dementia (FTD) Patients
Brief Title: Efficacy and Tolerability of Memantine in Frontotemporal Dementia (FTD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRD 05/1-E
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2005-01

CONDITIONS: Dementia
Keywords: frontotemporal dementia; Mémantine; Patients with frontotemporal dementia
MeSH Terms: conditions — Dementia; Frontotemporal Dementia | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: memantine

SUMMARY:
The purpose of this trial is to assess the efficacy and tolerability of memantine (anti-excitotoxic, neuroprotective treatment currently used in Alzheimer's disease [AD]) in frontotemporal dementia patients after a one-year treatment.

DETAILED DESCRIPTION:
Background: Frontotemporal dementia (FTD) is the first cause of dementia in the presenium (onset before the age of 65 years). Characterized by behavioral disorders, it is often more incapacitating than Alzheimer's disease (AD), and leads to death within 7 years on average (9-10 years for AD). It affects young individuals (on average, 20 years younger than in AD), who are often still active. Management of these patients is therefore burdensome and complex. As opposed to AD, however, no treatment is currently available. Few therapeutic trials have actually been conducted on this disorder. Many reasons may account for this:

1. recent availability of reliable diagnostic criteria (the Lund and Manchester groups' consensus statement in 1994; revised in 1998),
2. the very small number of cases as opposed to AD-the number of cases was estimated at approximately 3,500 vs 600,000, for AD, in France in 2004-, FTD therefore falls into the category of rare diseases (i.e., less than 30,000 cases),
3. the scarcity of valuable physiopathological hypotheses.

Besides a non-specific serotoninergic dysfunction, no significant anomalies related to particular neuromediators have apparently been found (as opposed to AD, which is characterized by a cholinergic deficit). In 1998, the discovery of mutations in the Tau gene in certain kindreds showing a dominant autosomal transmission of FTD, oriented research efforts toward the tau protein and provided new perspectives. Many studies have suggested the role of excitotoxicity. Abnormal aggregation of the tau protein has been observed in the brains of a majority of FTD patients (familial and sporadic form). Excitotoxicity may be responsible for promoting this abnormal aggregation through modification of the expression and phosphorylation state of the tau protein. The hypothesis of this study is that an anti-excitotoxic neuroprotective treatment may slow the pathogenic process and therefore be an effective treatment for this pathology.

Goals: To assess the efficacy and tolerability of memantine (anti-excitotoxic, neuroprotective treatment currently used in AD) in FTD patients after a one-year treatment.

Type of study: National, multicenter, randomized, double-blind, parallel group, placebo-controlled, phase II therapeutic trial.

Study design: Sixty four (64) patients, aged 45 to 75 years, will be enrolled in the study for a period of 12 months (clinical inclusion criteria are defined based on the Lund and Manchester group consensus statement [revised version 1998]), and followed up for 1 year in a controlled study. At the time of inclusion, the Mini Mental Status Examination (MMSE) score should be at least 19 (below 18, a neuropsychological examination is impossible). Patients will either take memantine, or a placebo (randomization ratio of 1:1) twice a day (i.e., 20 mg of memantine per day in the memantine arm). The primary efficacy variable will be a global assessment tool, the CIBIC-Plus (Clinician's Interview-Based Impression of Change Plus Caregiver Input). Secondary efficacy variables will include behavioral scales [the NeuroPsychiatric Inventory (NPI), the Frontal Behavior Inventory (FBI)], cognitive scales [the Mattis Dementia Rating Scale (MDRS), the MMSE], activities of daily living (Disability Assessment for Dementia, DAD), time spent by the caregiver of the patient (Resource Utilization in Dementia, RUD), and caregiver burden scale (Zarit Burden Inventory), and tolerability of the drug. The main analysis will be carried out on an intention-to-treat basis in all randomized patients having undergone at least one evaluation after inclusion (the Last Observation Carried Forward LOCF value, will be attributed to missing values). This analysis will be carried out at the end of the double-blind study (main judgement criterion)

Expected results and perspectives: The main expected result is the confirmation of the efficacy of memantine as a treatment for FTD, which would set a precedent in the treatment of this disease. Such a result could also lead the way to the development of treatments for other related neurodegenerative disorders (tauopathies) such as the other frontotemporal lobar degenerations (semantic dementia, progressive non-fluent aphasia), progressive supranuclear palsy, or corticobasal degeneration. Finally, the standardized follow-up of a 64 patient cohort in this study will provide important information on the natural history of a rare and poorly-known disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FTD based on the criteria defined by the Lund and Manchester groups' consensus statement (revised in 1998), whose disease has been progressing during the last year.
* MMSE score of 19 or higher
* Men and women aged 45 to 75 years
* Without speech, visuospatial, or episodic memory impairments

Exclusion Criteria:

* Age > 76 years
* Illiterate or misunderstanding patients
* Patients with cancer, heart disease, lung disease, kidney disease (creatinine > 200 mg/dL), or epilepsy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Martine Vercelletto, MD, Study Director — Centre de la Mémoire, Clinique Neurologique CHU Nord Nantes 44093 France; mvercelletto@chu-nantes.fr; Lucette Lacomblez, MD, Principal Investigator — Federation de Neurologie AP-HP Paris 75 013 France; lucette.lacomblez@psl.ap-hop-paris.fr; Bruno Dubois, MD, Principal Investigator — Centre du Langage et de Neuropsychologie AP-HP Paris 75013 France; b.dubois@psl.ap-hop-paris.fr; Anne Sophie Rigaud, MD, Principal Investigator — Hôpital Broca, Paris 75 France; anne-sophie.rigaud@brc.ap-hop-paris.fr; Jean-Francois Dartigues, MD, Principal Investigator — Hôpital Pellegrin Bordeaux 33 076 France; jean-francois.dartigues@u.bordeaux2.fr; Sophie Auriacombe, MD, Principal Investigator — Hôpital Pellegrin Bordeaux 33 076 France ; sophie.auriacombe@u.bordeaux.fr; Philippe Couratier, MD, Principal Investigator — Hôpital Dupuytren, Limoges 87000 France; philippe.couratier@unilim.fr; Jacques Touchon, MD, Principal Investigator — Hôpital Gui de Chaulliac, Montpellier 34 295 France; jacques.touchon@wanadoo.fr; Matthieu Ceccaldi, MD, Principal Investigator — Hôpital de la Timone Marseille 13 005 France; mceccaldi@ap-hm.fr; Mira Didic, MD, Principal Investigator — Hôpital de la Timone Marseille 13005 France; mira.didic@medecine.univ-mrs.fr; Serge Bakchine, MD, Principal Investigator — Hôpital Maison Blanche, Reims 51 092 France; sbakchine@chu-reims.fr; Bernard-Francois Michel, MD, Principal Investigator — Hôpital Sainte Marguerite, 13009 France; bmichel@ap-hm.fr; Catherine Thomas-Anterion, MD, Principal Investigator — Hôpital Bellevue Saint Etienne, 42 000 France; catherine.thomas@chu-st-etienne.fr; Bernard Laurent, MD, Principal Investigator — Hôpital Bellevue Saint Etienne 42 000 France; bernard.laurent@univ-st-etienne.fr; Francois Sellal, MD, Principal Investigator — Hôpital Civil Strasbourg 67000 France; francois.sellal@chru-strasbourg.fr; Serge Belliard, MD, Principal Investigator — Hôpital Pontchaillou Rennes 35 000, France; serge.belliard@chu-rennes.fr; Herve Allain, MD, Principal Investigator — Service de Pharmacologie, CHU de Rennes 35 000 France ; Herve.allain@univ-rennes1.fr; Michele Puel, MD, Principal Investigator — Hôpital Purpan, Toulouse 31059 France; PUEL.M@chu-toulouse.fr; Jean-Francois Demonet, MD, Principal Investigator — Clinique Neurologique CHU Purpan Toulouse 31059 France; demonet@toulouse.inserm.fr; Marie Sarazin, MD, Principal Investigator — Centre du Langage et de la Mémoire, Hôpital de la Salpétriére AP-HP Paris 75013 France
Locations (1):
- Martine Vercelletto, Nantes, France

REFERENCES:
- [Derived] Boutoleau-Bretonniere C, Lebouvier T, Volteau C, Jaulin P, Lacomblez L, Damier P, Thomas-Anterion C, Vercelletto M. Prospective evaluation of behavioral scales in the behavioral variant of frontotemporal dementia. Dement Geriatr Cogn Disord. 2012;34(2):75-82. doi: 10.1159/000341784. Epub 2012 Aug 23. PMID 22922703
- [Derived] Vercelletto M, Boutoleau-Bretonniere C, Volteau C, Puel M, Auriacombe S, Sarazin M, Michel BF, Couratier P, Thomas-Anterion C, Verpillat P, Gabelle A, Golfier V, Cerato E, Lacomblez L; French research network on Frontotemporal dementia. Memantine in behavioral variant frontotemporal dementia: negative results. J Alzheimers Dis. 2011;23(4):749-59. doi: 10.3233/JAD-2010-101632. PMID 21157021